CLINICAL TRIAL: NCT03929432
Title: Treatment Outcomes and Brain Mechanisms Associated With Non-Invasive Neuromodulation in Post-Stroke Aphasia
Brief Title: Treatment Outcomes With tDCS in Post-Stroke Aphasia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Arkansas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 207342
Record Dates: First submitted 2019-04-15; First posted 2019-04-26 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Aphasia
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Active tDCS versus sham tDCS will be masked to the participants
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active tDCS (with Speech-Language Treatment) (Active Comparator): tDCS Stimulation Dose: 1.5 mA for 20-mins
  Interventions: Device: Active Transcranial Direct Current Stimulation with SLT
- Sham tDCS (with Speech-Language Treatment) (Sham Comparator): No tDCS stimulation
  Interventions: Device: Sham Transcranial Direct Current Stimulation with SLT

INTERVENTIONS:
Device: Active Transcranial Direct Current Stimulation with SLT — Soterix Medical 1×1 transcranial Direct Current Stimulator for Clinical Trials (1x1 tDCS-CT).
  Excitatory stimulation to the left hemisphere will be achieved through a 1x1 montage utilizing two carbon-rubber electrodes and 5x7 EASY pad sponges (A-tDCS [excitatory]left target; C-tDCS [inhibitory]right hemisphere). Each PWA will have a unique 5-digit tDCS program code for each treatment phase. One code will instruct the 1x1 tDCS-CT to administer active stimulation as describe above (i.e., 1.5 mA for 20 min). The other will administer 1.5 mA for only a few seconds to simulate active stimulation. SLT will consist of Semantic Feature Analysis, Phonological Component Analysis, and Verb Network Strengthening Treatment
  Arms: Active tDCS (with Speech-Language Treatment)
Device: Sham Transcranial Direct Current Stimulation with SLT — Control condition in which only SLT is administered.Participant receives 1.5 mA for only a few seconds to simulate active stimulation, then the stimulation will cease. SLT will consist of Semantic Feature Analysis, Phonological Component Analysis, and Verb Network Strengthening Treatment
  Arms: Sham tDCS (with Speech-Language Treatment)

SUMMARY:
The purpose this study is to test the utility of pairing external neuromodulation with behavioral language treatment to boost therapy outcomes and to investigate the mechanisms associated with recovery. Because all PWA have word retrieval deficits, this project will test if greater language gains can be achieved by supplementing anomia intervention with excitatory brain stimulation to the left hemisphere and will evaluate associated functional brain changes to aid the optimization of neural reorganization to facilitate language processing.

DETAILED DESCRIPTION:
Aphasia is a language impairment that commonly occurs following brain damage (e.g., stroke). While language rehabilitation can yield improved language functioning, treatment outcomes vary greatly across individuals. In chronic aphasia, language gains occur through the brain's inherent ability to reorganize (i.e., neuroplasticity).

While Speech-language therapy (SLT) can target various language skills and modalities, the most pervasive deficit across all persons with aphasia (PWA) is difficulty with word finding. Thus, aphasia treatment often includes some form of intervention focused on improving naming abilities. As with language function in general, naming abilities in PWA seems to be associated with left hemisphere recruitment, particularly with the viable tissue at the rim of the lesion (perilesional areas). This project investigates an innovative approach to improving current therapy by examining the benefits of using excitatory transcranial direct current stimulation (tDCS) stimulation/neuromodulation during anomia treatment (i.e. word-finding treatment).

This study investigates an innovative approach to improving current therapy by examining the benefits of using excitatory tDCS stimulation/neuromodulation during anomia treatment. This project will provide novel mechanistic understanding of changes in functional brain connectivity in persons with post-stroke aphasia and how connectivity relates to treatment outcomes.

The aims of this study are as follows:

Aim 1. To investigate the benefits of using broad transcranial direct current stimulation (tDCS) to improve word retrieval in persons with aphasia (PWA). Aim 2. To study functional brain changes related to this treatment. Aim 3. To examine behavioral and neural re-organization correlates related to treatment outcomes.

All participants will complete the following 3 components: (1) Baseline Assessment, (2) Interventions (i.e., SLT with active tDCS & sham tDCS , and (3) Outcome Testing (i.e., Behavioral & Brain Imaging). During the first week, each participant will complete all of the Neuropsychological Testing Battery and the first round of the outcome measures as pre-testing before starting SLT. Then the participant will complete 2 weeks of SLT accompanied with either active tDCS or sham tDCS. Once the SLT is completed, the participant will complete round 2 of outcome testing (i.e., post-testing for 1st SLT phase and pre-testing for 2nd SLT phase). Then, the participant will complete another 2 weeks of SLT but with the other tDCS condition. Once SLT is completed, the participant will complete round 3 of outcome testing (i.e., post-testing for 2nd SLT phase). Lastly, the participant will complete round 4 of outcome testing (i.e., follow-up)

ELIGIBILITY:
Inclusion Criteria:

* Presence of post-stroke aphasia
* Single left hemisphere stroke etiology
* At least 6 months post-stroke
* Age range between 18 and 80 years old
* Speak English as a native language
* Adequate hearing and vision to complete the tasks

Exclusion Criteria:

* Severe auditory comprehension deficits (determined by pretest) (i.e., global aphasia, Wernicke's aphasia, transcortical sensory aphasia)
* Inability to provide informed consent
* Co-occurring history of neurological disease/disorder/injury (e.g., traumatic brain injury, right hemisphere stroke, dementia)
* Co-occurring history of a major mental illness (e.g., schizophrenia, drug addiction, bipolar)
* Clinical conditions contraindicated for MRI or tDCS (e.g., implanted electrical devices, claustrophobia, seizure disorder)
* Positive pregnancy test (for females)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-09-03 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Change in correct naming of nouns on Philadelphia Naming Test. | Immediately after 1st and 2nd treatment phases and at 10 follow up after study completion
  Naming gains for untreated items.

SECONDARY OUTCOMES:
Change in correct naming of verbs on Action Naming Test | Immediately after 1st and 2nd treatment phases and at 10 follow up after study completion
  Naming gains for untreated items.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Moser, PhD, CCC-SLP, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

IPD SHARING:
Plan to Share IPD: No